CLINICAL TRIAL: NCT02513888
Title: Prevention of Type 2 Diabetes in Women With Prediabetes Using Vitamin D Supplementation and Lifestyle Intervention in North India (PREVENT-WIN Study)
Brief Title: Prevention of Type 2 Diabetes With Vitamin D Supplementation
Acronym: PREVENT-WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, Dr Anoop Misra, Investigator, Diabetes Foundation, India
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: PREVENT_WIN_RURAL
Record Dates: First submitted 2015-07-29; First posted 2015-08-03 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2018-07

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Vitamin D; Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D + diet and lifestyle (Experimental): subjects will be given vitamin D supplement will be given along with diet nd lifestyle modification
  Interventions: Dietary Supplement: vitamin D + diet and lifestyle
- placebo + diet and lifestyle (Placebo Comparator): Subjects will be given placebo with diet and lifestyle
  Interventions: Dietary Supplement: Placebo + diet and lifestyle

INTERVENTIONS:
Dietary Supplement: vitamin D + diet and lifestyle — subjects will be given vitamin D along with diet and lifestyle modification counselling
  Arms: Vitamin D + diet and lifestyle
Dietary Supplement: Placebo + diet and lifestyle — placebo along with diet and lifestyle modification counselling
  Arms: placebo + diet and lifestyle

SUMMARY:
PREVENT-WIN study has three components.

The work plan will have the following S&T components. Component 1: Cross-sectional Study

Cross-sectional study will be of 1.5 years where 400 women from rural will be screened randomly for the vitamin D deficiency and its determinants including duration of sun exposure.

Component 2: Prospective Study

This open-label randomized placebo-controlled trial would be done in 150 pre-diabetic women with vitamin D deficiency. The women will be recruited from cross-sectional study, out patient department and health camps and they will be followed up for 2 years. The women will be randomized into two groups; lifestyle modification counseling along with intervention with either vitamin D or placebo. The levels of vitamin D and blood glucose will be assessed periodically (every 6 months). In those having recurrent vitamin D deficiency, the course of vitamin D will be repeated. At the end of the study, incidence of T2DM in both groups will be compared.

Component 3: Information Education and Communication (IEC) Activities:

There is a paucity of IEC material on vitamin D deficiency in women residing in rural areas. IEC material will be developed and IEC activities through various modes like lectures, workshops, group discussions, leaflets/booklets distribution and audio video media shows (Hindi and English) will be used for educating health professionals, Medical and paramedical workers and various village level health functionaries like, Multi purpose workers, anganwadi workers, Accredited Social Health Activist under National Rural Health Mission of Government of India (ASHA). Besides this, Self Help Groups (SHGs) and women will be told about the benefits of balance diet, dietary intake of calcium, vitamin D, benefits of sun exposure and adverse health effects of vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* 1. Prediabetes:

  1. Fasting blood glucose ≥100mg/dl and <126mg/dl, or
  2. 2-h plasma glucose ≥140mg/dl and <200mg/dl (after ingestion of 75 g anhydrous oral glucose), and 2. Baseline level of 25 hydroxy vitamin D <30ng/dl. 3. Women aged 20-60 years

Exclusion Criteria:

1. Received Vitamin D and/or calcium supplementation in the previous six months.
2. On any medication within last one month which could potentially influence insulin secretion, insulin sensitivity, vitamin D or calcium metabolism (eg metformin, thiazolidione, steroids etc) and on any medication that activate steroid and xenobiotic receptor and drugs used in transplantation (e.g. steriods, calcitonin etc.)
3. Pregnancy and lactation at the time of study.
4. Severe end organ damage or chronic diseases: renal/ hepatic failure, any malignancy, nephrotic syndrome, malabsorption etc.
5. Known case of HIV infection.
6. Primary or tertiary hyperparathyroidism, granulomatous disorders (e.g. sarcoidosis) and any lymphomas
7. Known case of diabetes mellitus. -

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
fasting glucose (mg/dL) | 2 years

SECONDARY OUTCOMES:
TC (mg/dL) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Puneet Misra, MD, Principal Investigator — All India Institute of Medical Sciences, New Delhi, India
Locations (1):
- Comprehensive Rural Health Services Project, AIIMS, Ballabgarh, Haryana, India

REFERENCES:
- [Derived] Misra P, Kant S, Misra A, Jha S, Kardam P, Thakur N, Bhatt SP. A Community Based Randomized Controlled Trial to See the Effect of Vitamin D Supplementation on Development of Diabetes Among Women with Prediabetes Residing in A Rural Community of Northern India. J Family Med Prim Care. 2021 Aug;10(8):3122-3129. doi: 10.4103/jfmpc.jfmpc_311_21. Epub 2021 Aug 27. PMID 34660457